CLINICAL TRIAL: NCT06059794
Title: Assessment of Anxiety Disorder in Relation to PUQE Score of Nausea and Vomiting in First Trimester Pregnancy
Brief Title: Anxiety in Relation to Nausea and Vomiting in Pregnancy
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, principal investigator, Ain Shams Maternity Hospital
Other Study IDs: FMASU MS 717/2022
Record Dates: First submitted 2023-09-16; First posted 2023-09-29 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Nausea Gravidarum; Anxiety
Keywords: PUQE score; GAD-7 questionnaire
MeSH Terms: conditions — Anxiety Disorders | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PUQE score — The Pregnancy-Unique Quantification of Emesis (PUQE) is a scoring system to quantify the severity of nausea and vomiting of pregnancy (NVP). Based on quantification of the 3 physical symptoms of NVP (nausea, vomiting and retching)
Other: GAD-7 — The Generalised Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day"

SUMMARY:
The goal of this observational study is to learn more about the relation between anxiety (assessed by GAD-7 questionnaire) and the nausea and vomiting in pregnancy (objectively measured by PUQE score).

Participants will answer 2 questionnaires: (GAD-7) for anxiety; and (PUQE score) for nausea and vomiting.

DETAILED DESCRIPTION:
Study Procedures:

* Protocol approval will be sought from the ethical committee of the department of Obstetrics & Gynecology, Faculty of Medicine, Ain Shams University.
* Recruitment of pregnant women complaining of nausea and vomiting in pregnancy (NVP) in first trimester will be done from the outpatient clinic and antenatal ward in Ain Shams University Maternity Hospital.
* An informed written consent will be taken from all participants before enrollment in the study.
* History taking, examination, and investigations (CBC, ultrasound, acetone in urine, serum sodium, potassium, alanine transaminase (ALT), aspartate transaminase (AST), serum creatinine) will be done to identify eligible patients according to the inclusion and exclusion criteria.
* PUQE score will be calculated for each patient. Patients will be classified into 3 groups (mild, moderate, severe) accordingly.
* GAD-7 questionnaire will be calculated for each patient. Degree of anxiety will be classified into 4 groups (minimal, mild, moderate, severe) accordingly.
* Data will be recorded in a case report form.
* Statistical analysis will be done accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in first trimester complaining of NVP
* Age (18-40) years

Exclusion Criteria:

* History of known medical problem (e.g., endocrine abnormalities, gastrointestinal disease).
* Known current or past psychiatric disorder (e.g., depression, anxiety, bipolar disorder, delirium, eating disorders, and psychotic disorder)
* Multiple pregnancy
* Known obstetric complications (non-viable pregnancy; either ectopic pregnancy; gestational trophoblastic disease, or miscarriage).
* Medications (including antidepressant, anti-psychotic or other psychiatric drugs during the last 6 months) or illegal drug or narcotic use that would affect the test results
* Current or past history of cognitive incompetence which can make it difficult to understand how to score GAD-7 questionnaire.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: the study will include 105 pregnant women recruited from antenatal clinic and antenatal ward
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Pregnancy-Unique Quantification of Emesis (PUQE) score | Baseline
  The Pregnancy-Unique Quantification of Emesis (PUQE) is a scoring system to quantify the severity of nausea and vomiting of pregnancy, based on quantification of the 3 physical symptoms of (nausea, vomiting and retching).
Generalised Anxiety Disorder Assessment (GAD-7) | Baseline
  The Generalised Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day"

SECONDARY OUTCOMES:
Disturbance in Sodium. | immediately after the intervention
  assessed by serum levels of Sodium.
Disturbance in Potassium | immediately after the intervention
  assessed by serum levels of Potassium.
Dehydration | immediately after the intervention
  dehydration as detected clinically (like oliguria)
Ketonuria | immediately after the intervention
  acetone in urine assessed by urine dipstick
Hospital admission | immediately after the intervention
  Hospital admission
Hospital stay | immediately after the intervention
  Duration of hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Khaled IA Abdalla, MD, Study Chair — Ain Shams University; Ebtihal M El Taieb, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol and analytic code will be shared after completion and publication of the study
Supporting Information: Study Protocol, Analytic Code
Time Frame: For 2 years after completion and publication of the study
Access Criteria: An email will be sent upon reasonable request